CLINICAL TRIAL: NCT05405400
Title: Understanding Longer-term Effects of a Father-engaged, Play-based Home Visiting Intervention to Promote Early Childhood Development and Prevent Violence in Rwanda: The Sugira Muryango Longitudinal & Spillover Study
Brief Title: The Sugira Muryango Longitudinal & Spillover Study
Status: Completed | Type: Observational
Sponsor: Boston College (Other)
Collaborators: University of Rwanda (Other); FXB-Rwanda (Unknown); LEGO Foundation (Unknown); The ELMA Foundation (Other); Echidna Giving (Unknown); Wellspring Philanthropic Fund (Unknown); United States Agency for International Development (USAID) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Theresa Betancourt, Salem Professor in Global Practice, Boston College
Other Study IDs: 22.198.01
Record Dates: First submitted 2022-05-27; First posted 2022-06-06 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-08

CONDITIONS: Cognitive Change; Growth; Stunting, Nutritional; Language; Depression; Behavior; Violence; Parenting
Keywords: Early childhood development; Intimate partner violence; Rwanda; Intervention; Longitudinal
MeSH Terms: conditions — Growth Disorders; Language; Depression; Behavior

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Treatment group: Families in the treatment group received one welcome visit, 12 visits from a community-based volunteer trained in the Sugira Muryango intervention over 3-4 months, as well as booster visits at 3 and 6 months. The primary caregiver, secondary caregiver if applicable, and any children ages 6-36 months participated in the sessions. Other family members were welcome to join as available.
- Control group: Usual childcare (no intervention)

SUMMARY:
The Early Childhood version of Sugira Muryango is a family-based, home-visiting intervention targeted at early childhood development and implemented with families living in extreme poverty in three districts of Rwanda. This version of Sugira Muryango was first tested in two small pilot studies and a large cluster randomized trial (CRT) was implemented between February 2018 and September 2019 . Pre- to post-intervention findings demonstrated that Sugira Muryango led to improvements in caregiver behaviors linked to child development and health as well as reductions in violence, which were sustained 12 months after the intervention, at which time improvements in child development were observed.

The Research Program on Children and Adversity in the Boston College School of Social Work is led by Dr. Theresa S. Betancourt and will, in partnership with the University of Rwanda, FXB-Rwanda and Laterite, conduct a longitudinal follow-up study to investigate the longer-term outcomes of the Sugira Muryango intervention in families who participated in the CRT. The four-year follow-up will examine the long-term and sustained outcomes of the intervention. In particular, the investigators will look at key indicators of long-term positive outcomes for children such as school readiness and transition to formal schooling. Given the lack of longitudinal research on intervention programs supporting ECD in sub-Saharan Africa, this study will contribute greatly to the body of knowledge on the costs and benefits of investments in ECD and guide policy makers and government leaders on making impactful investments in children, leading to long-term benefits for the population at large.

The follow-up study involves two activities:

Activity A: Pilot to assess measures performance of newly added measures and field test study protocols.

Activity B: Four-year follow-up of families who participated in the CRT of the Sugira Muryango intervention.

DETAILED DESCRIPTION:
The aim of the study is to assess the impacts of Sugira Muryango on treated families compared to families receiving only usual care (controls) four years after the intervention. Moreover, at this visit, the investigators will also for the first time examine potential spillover effects of Sugira Muryango onto siblings of children enrolled in the original study. The longitudinal follow-up study will assess whether and to what extent Sugira Muryango has an impact on caregivers' awareness and utilization of available services; support for children's education and playful learning; home hygiene; parenting practices, including child feeding/nutrition, stimulation and sensitive care; experiences of intimate partner violence; use of harsh discipline; mental health, including depression and alcohol use; gender attitudes; and overall wellbeing. It will also assess whether and to what extent Sugira Muryango has an impact on children's physical development; cognitive and linguistic development; temperament; enrollment in early or formal education; school readiness, including self-regulation and early literacy and numeracy; mental health, including internalizing and externalizing and depression; behavior, including conduct problems; and gender attitudes. Finally, the study will assess potential covariates such as the impact of the COVID-19 pandemic and associated lockdowns, child disability, and household size and composition.

The specific objectives are:

To assess the long-term (4 years post-intervention) impact of Sugira Muryango on caregiver behaviors, attitudes, mental health and wellbeing, especially as related to parenting and intimate partner violence.

To assess the long-term (4 years post-intervention) impact of Sugira Muryango on previously enrolled children's physical and cognitive development and health.

To assess the long-term (4 years post-intervention) impact of Sugira Muryango on previously enrolled children's behavior, mental health, school readiness and gender attitudes.

To assess the long-term (4 years post-intervention) impact of Sugira Muryango on younger and older siblings of children enrolled in the intervention, including on their physical and cognitive development and health, and in the case of older siblings their school readiness, behavior and gender attitudes.

The following activities will be conducted during the proposed 4-year follow up study:

* Activity A: Pilot to assess measures performance and field test study protocols.

  * Phase A1: Translation and adaptation of newly selected measures.
  * Phase A2: A Pilot study of selected new child measures with 150 children and their primary caregivers in a sector of the Sugira Muryango PLAY Collaborative Expansion Study to test the feasibility and validity of new tools.
* Activity B: Four-year follow-up of families who participated in the Cluster Randomized Trial (CRT) of the Sugira Muryango intervention.

  * Phase B1: Household tracking and re-enrollment of 1,049 households that participated in the prior CRT (April-May 2022).
  * Phase B2: Quantitative (full sample) and qualitative (subsample) data collection with the 1,049 households from the prior CRT, including children and caregivers who were in the original CRT, and siblings in a subset of households to test for spillover effects (June [Quantitative] & December [Qualitative] 2022).

Our specific hypotheses are as follows:

Longitudinal Hypotheses

1. Sugira Muryango will have effects (superior when compared to usual care households) on a range of outcome domains, both new domains and those assessed in the prior CRT.

   1. Sugira Muryango will continue to have effects among eligible caregivers and children compared to controls on a range of outcomes assessed at previous waves of data collection, and
   2. Sugira Muryango will have effects on new outcomes that have become relevant as the children have aged, including aspects of school readiness.

   Spillover Hypothesis
2. Sugira Muryango will have positive effects on younger and older siblings of children who were eligible for and participated in the intervention compared to siblings in usual care households.

Secondary exploratory analyses Analyses evaluating potential child and caregiver sex differences will be performed across all outcomes to examine differences in parenting behaviors and child outcomes as children get older and approach school age.

Study benefits and justification Potential societal benefits of the study include increased knowledge about evaluating ECD and parenting in Rwanda, increased knowledge of ECD in Rwanda, and increased knowledge regarding family-based ECD interventions to improve child development outcomes in low-resource settings. Intervening in early childhood has been demonstrated to be highly cost-effective for improving child development and life outcomes, yet interventions in low-resource settings-particularly in sub-Saharan Africa-are limited and not always well-evaluated or systematically implemented. At the individual level, families who participate in the study will receive free disability and behavioral screening for eligible children and will be connected with support services should a disability or other risk of harm be identified.

The key research question is whether Sugira Muryango provides lasting benefits to children in households that received the intervention. Little longitudinal research into home-visiting ECD interventions in this region exists; findings from the proposed research will add critical evidence to inform Rwanda's expansion of ECD support to families as well as learnings for other countries.

The study has been reviewed and approved by the Rwanda National Ethics Committee, the National Institute of Statistics of Rwanda, and the National Council for Science and Technology in Rwanda.

ELIGIBILITY:
Participated in the Sugira Muryango CRT in 2018-19 (Trial Registration Number NCT02510313).

Family inclusion criteria for the CRT were:

* living in the Rubavu, Ngoma or Nyanza District of Rwanda
* being VUP-eligible (according to the Rwandan government)
* having at least one child aged 6-36 months living in the home
* having at least one caregiver who was willing to discuss and enhance their caregiving practices by interacting with a home-visiting coach (a community-based volunteer or CBV).

Further caregiver inclusion criteria were:

* was aged 18 or older and cared for child(ren)
* lived in the same household as the child(ren). For the current Longitudinal Study, inclusion criteria for families are
* having participated in the prior CRT
* living in Ngoma, Nyanza, or Rubavu districts
* having at least one child who participated in the CRT and who is currently living in the household.

Inclusion criteria for younger siblings are:

* aged 3 months or older
* was not eligible to participate in the original CRT due to age (below 6 months or not yet born at the time of CRT).

Inclusion criteria for older siblings are:

* aged 12 years or younger
* lived in the household but was not eligible to participate in the original CRT due to age (above 36 months at the time of CRT)
* currently lives in the household that participated in the CRT.

Exclusion Criteria:

Other than not meeting inclusion criteria, specific family exclusion criteria for the CRT were:

* caregiver(s) having severe cognitive impairments which precluded their ability to speak to the research questions under study
* families or caregivers being in the midst of crisis (e.g., a caregiver(s) with active suicidal attempts or psychosis). Families with ongoing crises or disabilities were excluded from the study and were referred to appropriate services.
* These exclusion criteria remain the same for the current Longitudinal study.
* Siblings will be excluded from sampling for the spillover study if the primary caregiver has been away from the household for six months or more.

Min Age: 3 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The population consists of families who participated in the earlier CRT. Families for the CRT were randomly selected from government-provided lists of families who were eligible for the Vision Umurenge Program (VUP). Families' participation in the VUP and selection into one of two versions of the VUP program, namely classic public works (cPW) or expanded public works (ePW), was determined by governmental policies and was not under the control of the research team. Eligibility for VUP indicates that the family was in the poorest category under Rwanda's poverty categorization system (Ubudehe 1). Families were living in Ngoma, Nyanza or Rubavu district of Rwanda and had at least one child between the ages of 6-36 months.
Sampling Method: Probability Sample
Enrollment: 2932 (Actual)
Dates: Start 2022-04-20 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
"Home Observation Measurement of the Environment" infants/toddlers survey and early childhood survey | Through study completion (4 years)
  Observation of caregiver engagement and stimulation of children (younger siblings and CRT children)
"Ages & Stages Questionnaire - 3" | Through study completion (4 years)
  Caregiver report on child's development (younger siblings)
"Mullen Scale of Early Learning" | Through study completion (4 years)
  Observation of child's cognitive, motor, and linguistic development (younger siblings)
"Kaufman Assessment Battery for Children-2" | Through study completion (4 years)
  Observation of child's cognitive and linguistic development (CRT children and older siblings)
"Wechsler Preschool & Primary Scale of Intelligence" | Through study completion (4 years)
  Observation of child's cognitive and linguistic development
"International Development & Early Learning Assessment" stimulating care and play module | Through study completion (4 years)
  Caregiver report on playful parenting activities and childcare arrangement (for all children)
"Multiple Indicator Cluster Survey" child discipline module | Through study completion (4 years)
  Caregiver self-report of child discipline practices and behaviors (for all children)
Combined module based on "Multiple Indicator Cluster Survey" and "ISPCAN Child Abuse Screening Tool" | Through study completion (4 years)
  Child self-report of experiences of discipline and violence (older siblings)
DHS "Intimate Partner Violence" survey | Through study completion (4 years)
  Caregiver self-report on victimization and perpetration of intimate partner violence
"Child Behavior Checklist" | Through study completion (4 years)
  Caregiver report on child's internalizing and/or externalizing (CRT children and older siblings)

SECONDARY OUTCOMES:
"Observation of Mother-Child Interactions" | Through study completion (4 years)
  Observation of caregiver's sensitive care (younger siblings)
"The Role of Play in Children's Learning" | Through study completion (4 years)
  Caregiver self-report on play for children's learning and development
"Parental Acceptance-Rejection Questionnaire" | Through study completion (4 years)
  Caregiver self-report of stimulating care and play
DHS/Promundo "Father Engagement & Financial Decision-Making" survey | Through study completion (4 years)
  Caregiver self-report of financial decision making and father engagement in the family
"Gender Equitable Men" scale | Through study completion (4 years)
  Caregiver self-report of views of gender and masculinity
"Multiple Indicator Cluster Survey (5)" WASH module | Through study completion (4 years)
  Caregiver self-report of home sanitation & hygiene
World Health Organization "Infant and Young Child Feeding Practices" survey | Through study completion (4 years)
  Caregiver self-report of feeding practices
"Hopkins Symptom Checklist (25)" | Through study completion (4 years)
  Diagnostic tool for depression and anxiety in caregivers
"Enrollment in early education" survey | Through study completion (4 years)
  Caregiver report of child's enrollment in early education
"Child Enrollment in Formal Education" survey | Through study completion (4 years)
  Caregiver report of child's enrollment in formal education
"Service utilization" survey | Through study completion (4 years)
  Caregiver self-report on services utilized, e.g. government and non-governmental inputs and services
Anthropometric measures: height in centimeters | Through study completion (4 years)
  Measure of child height in centimeters (younger siblings and CRT children)
"Preschool Self-Regulation Assessment" | Through study completion (4 years)
  Caregiver report of child's self-regulation (CRT children)
"Infant Behavior Questionnaire" | Through study completion (4 years)
  Caregiver report of child's temperament (younger siblings)
"Early Childhood Behavior Questionnaire" | Through study completion (4 years)
  Caregiver report of child's temperament (younger siblings)
"Early Grade Reading Assessment" | Through study completion (4 years)
  Assessment of early literacy skills in children (older siblings)
"Center for Epidemiological Studies Depression Scale" | Through study completion (4 years)
  Diagnostic tool for depression in children (older siblings)
"Gender Equitable Men" scale | Through study completion (4 years)
  Child self-report of views of gender and masculinity (older siblings)
Anthropometric measures: weight in kilograms | Through study completion (4 years)
  Measure of child weight in kilograms (younger siblings and CRT children)
Anthropometric measures: standardized height-for-weight | Through study completion (4 years)
  Height and weight will be combined and the resulting scores standardized and reported as z-scores (younger siblings and CRT children)
Anthropometric measures: standardized height-for-age | Through study completion (4 years)
  Height and age will be combined and the resulting scores standardized and reported as z-scores (younger siblings and CRT children)
Anthropometric measures: middle upper arm circumference in centimeters | Through study completion (4 years)
  Measure of child circumference of middle upper arm in centimeters (younger siblings and CRT children)

OTHER OUTCOMES:
"International Development & Early Learning Assessment" parent attitudes module | Through study completion (4 years)
  Caregiver self-report of attitudes towards children's education
"International Development & Early Learning Assessment" parent expectations module | Through study completion (4 years)
  Caregiver self-report of expectations towards children's education
Epstein survey | Through study completion (4 years)
  Caregiver self-report of support for children's education
World Health Organization "Alcohol Use Disorders Identification Test (AUDIT)" | Through study completion (4 years)
  Caregiver self-report of alcohol use and/or abuse
"Flourishing Scale" | Through study completion (4 years)
  Caregiver self-report on quality of life
"Gender Equitable Men" norms scale | Through study completion (4 years)
  Caregiver self-report of perceived norms related to gender and masculinity
"Youth Conduct Problems Scale - Rwanda" | Through study completion (4 years)
  Child self-report of conduct problems (older siblings)

CONTACTS AND LOCATIONS:
Overall Officials: Theresa S Betancourt, ScD, MA, Principal Investigator — Boston College
Locations (3):
- Rwanda (3):
  - Homes and community buildings, Ngoma
  - Homes and community buildings, Nyanza
  - Homes and community buildings, Rubavu

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Barnhart, D. A., Farrar, J., Murray, S. M., Brennan, R. T., Antonaccio, C., Sezibera, V., Ingabire, C., Godfroid, K., Bazubagira, S., Uwimana, O., Kamurase, A., Yousafzai, A., Betancourt, T. (2020). Lay-worker delivered home promotes early childhood development and reduces violence in Rwanda; a randomized pilot. Journal of Child and Family Studies; 29, 1804-1817. https://doi.org/10.1007/s10826-020-01709-1
- [Background] Betancourt, T. S., Franchett, E., Kirk, C. M., Brennan, R. T., Rawlings, L., Wilson, B., ... & Ukundineza, C. (2018). Integrating social protection and early childhood development: open trial of a family home-visiting intervention, Sugira Muryango. Early Child Development and Care; 190(2), 219-235.
- [Background] Betancourt TS, Jensen SKG, Barnhart DA, Brennan RT, Murray SM, Yousafzai AK, Farrar J, Godfroid K, Bazubagira SM, Rawlings LB, Wilson B, Sezibera V, Kamurase A. Promoting parent-child relationships and preventing violence via home-visiting: a pre-post cluster randomised trial among Rwandan families linked to social protection programmes. BMC Public Health. 2020 May 6;20(1):621. doi: 10.1186/s12889-020-08693-7. PMID 32375840
- [Background] Britto PR, Lye SJ, Proulx K, Yousafzai AK, Matthews SG, Vaivada T, Perez-Escamilla R, Rao N, Ip P, Fernald LCH, MacMillan H, Hanson M, Wachs TD, Yao H, Yoshikawa H, Cerezo A, Leckman JF, Bhutta ZA; Early Childhood Development Interventions Review Group, for the Lancet Early Childhood Development Series Steering Committee. Nurturing care: promoting early childhood development. Lancet. 2017 Jan 7;389(10064):91-102. doi: 10.1016/S0140-6736(16)31390-3. Epub 2016 Oct 4. PMID 27717615
- [Background] Jensen SK, Placencio-Castro M, Murray SM, Brennan RT, Goshev S, Farrar J, Yousafzai A, Rawlings LB, Wilson B, Habyarimana E, Sezibera V, Betancourt TS. Effect of a home-visiting parenting program to promote early childhood development and prevent violence: a cluster-randomized trial in Rwanda. BMJ Glob Health. 2021 Jan;6(1):e003508. doi: 10.1136/bmjgh-2020-003508. PMID 33514591

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-05-25): https://cdn.clinicaltrials.gov/large-docs/00/NCT05405400/Prot_SAP_000.pdf